CLINICAL TRIAL: NCT05207293
Title: Pilot Test of Clinical Outcome Assessment Methodology (Primarily the Ordinal Scale of Clinical Improvement) and Other Symptom Assessment Patient-reported Outcomes Scales) and Qualitative Evidence of Content Validity
Brief Title: Pilot Test of COVID-19 Related Clinical Outcome Assessment Methodology and Qualitative Evidence of Content Validity
Status: Completed | Type: Observational
Sponsor: Synairgen Research Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: SG019
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; Ordinal Scale of Clinical Improvement; Clinical Outcome Assessment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is an acute respiratory disease caused by Severe Acute Respiratory Syndrome coronavirus (SARS-CoV).

Synairgen is currently conducting a global Phase III clinical trial of SNG001 to determine efficacy and safety in patients hospitalised due to COVID-19 that receive oxygen therapy. The primary endpoint in the Phase III trial (SG018) is to evaluate recovery in patients hospitalised due to COVID-19 that require oxygen therapy after administration of SNG001 compared to placebo. The primary endpoint will be determined using the World Health Organization Ordinal Scale of Clinical Improvement (OSCI) score, which will be assessed daily. The OSCI will be used in two different ways during SG018. When the patients are in hospital, the clinical study staff will assess the patient via observation using the OSCI. However, when patients have been discharged from hospital, the clinical study staff will assess the OSCI by asking two questions, one regarding the presence of COVID-19 symptoms and the other regarding usual activities returning to baseline levels. The patient will be required to answer both questions with either a 'yes' or 'no' answer. Daily assessments of the OSCI will be conducted via video call or telephone call after discharge from hospital. The two questions asked of patients when OSCI is assessed after discharge from hospital have been added to trial SG018 to allow assessment of OSCI to continue throughout the trial. As these are new questions and the data from these is being used to assess the primary endpoint in trial SG018, their relevance, ease of understanding and clarity needs to be shown, which is why this interview study is being conducted. Having patients comment on these questions will ensure that the way the benefit of treatment is being measured in SG018 is done in a robust and patient-centred way.

The main aims of this qualitative pilot study are to:

1. To confirm how relevant, clear and easy to understand the two additional OSCI questions asked about COVID-19 symptoms and levels of usual activity are when patients have been discharged from hospital.
2. To find out what other symptoms and experiences patients hospitalised for COVID-19 might have had to see if these are reflected in the questionnaires used in SG018.

DETAILED DESCRIPTION:
This is non-interventional, qualitative interview study. Patients will participate in a single one-on-one, semi-structured, 90-120 minute interview. The interviews will be audio/video-recorded. The interviews are non treatment-related, and no investigational drugs, devices, or invasive procedures will be administered or evaluated as part of this study.

Patients who have been hospitalized due to COVID-19 will be approached about the study by a dedicated clinician from the site the patient was hospitalized at. Eligible patients will be recruited via hospitals in the UK and the US. At that time, potential participants will be provided with the 'Consent to Contact' form, Patient Information Sheet and Informed Consent Form and if the patient is interested in the study the patient will be asked to sign 'Consent to Contact' form that will allow the clinical staff to pass the patient information to the research team at Parexel. All other research related activities will be conducted by the research team at Parexel.

Parexel research team will contact the potential participants to further confirm eligibility criteria, provide additional details of the study and explain the consent process. Participants will be given ample time to consider the study and the opportunity to ask the research team questions prior to deciding whether to participate or not.

If the participant agrees to take part in the study, the participant will be asked to provide signed consent by signing the Informed Consent Form.

Parexel research team will discuss the most suitable day and time for the interview and will assure that the participant has access to the required technology.

The interview is planned to last between 90-120 minutes and will be audio/video-recorded and transcribed to assure that all important information shared by the participants were captured and that data from the interview can be analysed in a qualitative manner with the use a qualitative data analysis software.

During the interview, the Parexel research team member with expertise in qualitative interviewing will conduct the interviews.

Before the interview begins, the interviewer will again explain the purpose of the study and the interview methodology to each participant. The semi-structured interviews will be conducted in four parts using a semi-structured interview guide.

The first part of the interview will include socio-demographic questions to collect data that can describe the participant interview sample. The following information will be collected: age, gender, nationality, place of residence, race, work status, level of education, general health status, chronic conditions, COVID-19 history including details regarding date of diagnosis, hospitalisation length, oxygenation, perception of COVID-19 severity.

The second part of the interview will be structured to evaluate the validity of the COVID-19 symptom assessment instrument and discharge OSCI via pilot study. Participants will first be asked to complete the instruments as would happen in the SG018 clinical trial. Participants will be asked to complete the PRO instrument using a think-aloud method, whereby participants are encouraged to verbalize their thoughts, while completing the instrument.

In the next step participants will be asked how relevant, clear and easy to understand these instruments were. Ease of completion, comprehensiveness, and appropriateness of the format, response scales, and recall period within the PRO instrument will be evaluated.

The last part of the interview will consist of the concept confirmation exercises where participants will be asked open-ended questions about their experience with COVID-19 to encourage spontaneous responses. This section of the interview guide will include topics, questions, and probes designed to evaluate the concepts collected via other PRO measures used in the Phase III study to confirm their acceptability. The topics covered will include patients' experience of COVID-19 symptoms, fatigue, signs of depression and anxiety, physical pain, impact on physical functioning and daily activities.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years at the time of consent
2. Must have a confirmed diagnosis of COVID-19
3. Must have been discharged from hospital due to COVID-19 infection in the last 35 days
4. Must exhibit reliability and physiologic capability (e.g. sufficient hearing, vision etc.) to comply with all protocol procedures, in the investigator's opinion and must have educational level of minimum 8th grade or primary school;

6. Must be able to read, write, and speak in a local language to complete the informed consent process and participate in an interview; 7. Must be willing to provide written informed consent to participate in the study; and, 8. Must be able to participate in a one-time interview for approximately 90-120 minute via video conference (e.g., Microsoft Teams, WebEx) AND has access to the necessary equipment and internet access.

Exclusion Criteria:

1. Signed the consent form to participate in the Synairgen SG018 clinical trial,
2. Cognitive impairment, significant mental illness, or other disability impairing ability to participate in and/or complete research interview based on study coordinator's or clinician's judgement; or,
3. Ongoing substance abuse disorders that may impact participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include up to 25 patients who have had a positive test for COVID-19 and who were hospitalised due to their COVID-19. Diagnosis of COVID-19 and hospitalization will be confirmed by study personnel. The interview will take place up to 35 days post discharge from hospital.
  The eligibility criteria are designed to align with the SG018 protocol to ensure that a similar population evaluates the PROs as the population who completes the instruments as part of the clinical development program.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Confirmation of content relevance, comprehensiveness and clarity | Within 35 days of hospital discharge
  Confirm the content relevance, comprehensiveness and clarity of the Ordinal Scale of Clinical Improvement (OSCI) score Patient Reported Outcome assessment post hospital discharge. Two questions are answered 'Yes' or 'No' and these determine a score of either 0, 1 or 2, where the higher the score the worse the outcome.
Confirmation of content relevance, comprehensiveness and clarity | Within 35 days of hospital discharge
  Confirm the content relevance, comprehensiveness and clarity of the COVID-19 symptom assessment instrument. When asked if the symptom is present, the patient answers either 'yes' or 'no'. The answer 'yes' indicates a worse outcome.
Confirmation of content relevance for SG018 PRO instruments (BCSS) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for the breathlessness, cough and sputum scale (BCSS) (scale of 0 (no symptoms) up to 4 (severe symptoms) to demonstrate the content relevance in this patient population.
Confirmation of content relevance for SG018 PRO instruments (EQ-5D-5L) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for EuroQol 5-dimension 5-level (EQ-5D-5L) to demonstrate the content relevance in this patient population. The EQ-5D-5L provides a simple descriptive profile and a single index value for health status. The EQ-5D-5L self-rated questionnaire includes a visual analogue scale, which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher health-related quality of life. It also includes the EQ-5D-5L descriptive system, which comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension. Here, 100 means the best health and 0 means the worst health.
Confirmation of content relevance for SG018 PRO instruments (GAD-7) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for the General Anxiety Disorder 7 Questionnaire (GAD-7) to demonstrate the content relevance in this patient population. Scoring will be done based on how often patients have been bothered by the problems as: feeling nervous, anxious or on edge; not being able to stop or control worrying; worrying too much about different things; trouble relaxing; being so restless that it's hard to sit still; becoming easily annoyed or irritable, and feeling afraid at if something awful might happen. The scores ranges from 0 to 4, where 0 represents not at all bothered by any of the above problems and 4 indicates nearly bothered every day by any of the above problems. Higher scores indicated worse outcome.
Confirmation of content relevance for SG018 PRO instruments (PHQ-9) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for the Patient Health Questionnaire-9 (PHQ-9) to demonstrate the content relevance in this patient population. Patient health questionnaire included: little interest or pleasure in doing things; feeling down, depressed or hopeless; trouble falling asleep or staying asleep, or sleeping too much; feeling tired or having little energy; poor appetite or overeating; feeling bad about yourself or that you are a failure have let yourself or your family down; trouble concentrating on things; moving or speaking so slowly or so fidgety or restless that you have been moving a lot more than usual; and thoughts that you would be better off dead; or thoughts of hurting yourself in some way. Based on responses, scoring will be done and scores ranges from 0 to 4, where 0 represents not at all bothered by any of the above problems and 4 indicates nearly bothered every day by any of the above problems. Higher scores indicated worse outcome.
Confirmation of content relevance for SG018 PRO instruments (FACIT) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for the FACIT Fatigue Scale (Version 4) (FACIT) to demonstrate the content relevance in this patient population. The FACIT Fatigue Scale (Version 4) will include statements for patients such as: I feel fatigued; I feel weak all over; I feel listless ("washed out"); I feel tired; I have trouble starting things because I am tired; I have trouble finishing things because I am tired; I have energy; I am able to do my usual activities; I need to sleep during the day; I am too tired to eat; I need help doing my usual activities; and I am frustrated by being too tired to do the things I want to do. Based on responses on above statements, scoring will be done and scores ranges from 0 to 4, where 0 represents not at all bothered by any of the above problems and 4 indicates very much bothered every day by any of the above problems. Higher scores indicated worse outcome.
Confirmation of content relevance for SG018 PRO instruments (BPI-SF) | Within 35 days of hospital discharge
  Conduct concept confirmation exercises for the Brief Pain Inventory (Short Form) (BPI-SF) to demonstrate the content relevance in this patient population. Form includes: did patient have pain other than everyday kinds of pain on assessment day; body part where patient feels pain; rate pain: at worst, at least in the last 24 hours, at average and at right now, by giving scores from 0 to 10, where 0 indicates no pain and 10 represents pain as bad as one can imagine; treatments or medications receiving for pain by patients; how much relief have pain treatments provided from 0% to 100%, where 0% represents no relief and 100% indicates complete relief; assessment of interference of pain in patients activity: general activity; mood; walking ability; normal work; relations with other people; sleep; enjoyment of life, and assessment will be done by scoring ranges from 0 to 10, where 0 represents pain does not interfere and 10 indicates pain completely interferes.

CONTACTS AND LOCATIONS:
Locations (5):
- Henry Ford Health System, Detroit, Michigan, United States
- United Kingdom (4):
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth, Dorset
  - Hull Royal Infirmary, Hull, East Riding Of Yorkshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Queen Elizabeth Hospital Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: Undecided